CLINICAL TRIAL: NCT02490254
Title: Childhood Uveitis Not Associated With Juvenile Idiopathic Arthritis: Incidence, Initial Management and One-year Outcomes
Brief Title: Childhood Uveitis Initial Management and One-year Outcomes
Status: Completed | Type: Observational
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: DALA1021
Record Dates: First submitted 2015-06-25; First posted 2015-07-03 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Any child (aged 0-16 years) with a new diagnosis of uni or bilateral uveitis.
  Interventions: Other: Surveillance card

INTERVENTIONS:
Other: Surveillance card

SUMMARY:
The investigators wish to establish a robust estimate of the incidence of inflammation inside the eye (uveitis) in children age 0-16 years in the UK, which hospitals children present to, where they are referred to, which treatment they receive during the first year after diagnosis, and how well they can see at the end of the first year.

DETAILED DESCRIPTION:
The investigators therefore propose to run a high quality surveillance study, together with the British Ophthalmological Surveillance Unit (BOSU) at the Royal College of Ophthalmologists and with the Scottish Ophthalmological Surveillance Unit (SOSU). BOSU and SOSU operate a monthly reporting card scheme. All UK consultant ophthalmologists and associate specialists receive a monthly 'report card' with a list of conditions being surveyed. Reporting clinicians will tick a box if they have seen a case of childhood uveitis in the preceding month, and return the card to BOSU/SOSU, who will inform us, the study investigators.

Following reporting of a new case, the investigators will directly contact reporting clinicians and send them a clinical proforma to collect clinical details about the case. At 12 months, a follow up questionnaire will be sent. The investigators will use only information available from patient case notes, with no direct patient contact. The investigators principal aim is to determine incidence of childhood uveitis in the UK. Secondary aims are to identify presentation patterns, referral pathways, associated medical conditions, management, and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Any child (aged 0-16 years) with a new diagnosis of uni or bilateral uveitis.

Exclusion Criteria:

* In England/Wales/Northern Ireland, children who are known to have pre existing juvenile idiopathic arthritis (joint inflammation) will be excluded. No exclusions will apply to the Scotland cohort.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Any child (aged 0-16 years) with a new diagnosis of uni or bilateral uveitis.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the total number of reported cases of uveitis. | 1 year
  A clinical proforma will be sent to the investigators collect clinical details about the case. At 12 months, a followup questionnaire will be sent.

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Dahlmann-Noor, Dr Med PhD, Principal Investigator — Moorfields Eye Hospital NHS Foundation Trust
Locations (1):
- Moorfields Eye Hospital NHS Foundation Trust, London, United Kingdom